CLINICAL TRIAL: NCT05953077
Title: The Effect of Prior Learning on Treatment of Morpheme Errors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DLD-Tx1
Record Dates: First submitted 2023-06-09; First posted 2023-07-19 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-01

CONDITIONS: Developmental Language Disorder
Keywords: treatment
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Intervention Model Description: quasi-experimental design with two active treatment groups
Who Masked: Care Provider
Masking Description: Parents are masked concerning children's specific language goals and treatment conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Easy first (Experimental): Children are treated for an emergent grammatical form that is used correctly at least 60% during three pre-treatment probe sessions. This form is treated until children generalize it's use an average of 90% or more across 3 probe sessions. Their treatment target is then switched to a grammatical form that is used less than 30% correct across 3 pre-treatment probe sessions.
  Interventions: Behavioral: Conversational recasting
- Hard first (Active Comparator): Children are treated for a grammatical form that is used accurately less than 30% of the time during 3 pre-treatment probe sessions. This form is treated until children generalize it's use an average of 90% or more across 3 probe sessions. Their treatment target is then switched to a grammatical form that is used less than 30% correct across 3 pre-treatment probe sessions.
  Interventions: Behavioral: Conversational recasting

INTERVENTIONS:
Behavioral: Conversational recasting — The treatment procedure uses 24 treatment doses embedded into child-friendly activities (crafts, book reading, play). Each each consists of a clinician eliciting use of a targeted grammatical form, a child's attempt (correct or incorrect) to use that form, and an immediate clinician repetition of the child's attempt (a recast), correcting any ungrammatical elements as needed. Clinicians must also attempt to gain the child's attention before providing the recast. Treatment sessions are approximately 30 minutes in duration.

SUMMARY:
This is a small-scale treatment study designed to determine which teaching methods result in the best learning. Treatment focuses on helping children with a developmental language disorder learn parts of grammar. Preschool children will receive assessments to determine whether they have a developmental language disorder and what parts of grammar they have not mastered. Children will receive one-on-one behavioral treatment over a six week period. Half of the children will be first taught a grammatical form they sometimes use and then one they rarely use. The other half will start with a grammatical form they rarely use. The study seeks to determine whether starting with something children sometimes use correctly (an easier part of speech) will speed later learning of something that is harder for them. The children's ability to use the grammatical forms taught to them will be assessed throughout the treatment period and approximately six weeks after treatment ends.

ELIGIBILITY:
Inclusion Criteria:

* Native English speaking
* Passed a pure-tone hearing screening
* 4-6 years of age
* SPELT-P2 (language) test score of < 87
* K-ABC-II Nonverbal Scale (cognition) test score of >75
* Sufficient morpheme errors to serve as treatment and control targets
* Articulations skills sufficient to judge use of language targets
* Able to attend treatment daily

Exclusion Criteria:

* Parent report of other handicapping conditions
* Clinical signs of other disorders
* Enrolled in outside treatment

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in the use of treated grammatical forms in untreated contexts | 3 days per week over 6 weeks
  Clinicians elicit ten uses of the trained grammatical form using toys, activities, and vocabulary with-held from treatment sessions. Change is assessed throughout the treatment period.
Change in the use of grammatical forms in untreated contexts | 3 days per week over 6 weeks
  Clinicians elicit ten uses of the untrained grammatical form using toys, activities, and vocabulary with-held from treatment sessions. Change is assessed throughout the treatment period.
Retention of trained grammatical forms | One session, approximately 6 weeks after treatment concludes.
  Clinicians elicit ten uses of the trained grammatical form using toys, activities, and vocabulary with-held from treatment sessions.
Retention of untrained grammatical forms | One session, approximately 6 weeks after treatment concludes.
  Clinicians elicit ten uses of the untrained grammatical form using toys, activities, and vocabulary with-held from treatment sessions.

SECONDARY OUTCOMES:
Change in spontaneous use | 5 sessions a week over 6 weeks.
  The number of unprompted use of the trained grammatical form that occurs during treatment sessions. Change is measured relative to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data, including clinical test scores and outcome measures, are shared in publications and presentations. Other study data is provided by request from the study PI.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Data is available for sharing after initial publication and for a minimum of 5 years after publication.
Access Criteria: Secondary use must be consistent with the intent of the original consent document.